CLINICAL TRIAL: NCT06788249
Title: Establishing Glutamatergic Changes as the Mechanism of Action in the Rapid Antidepressant Effects of Ketamine
Brief Title: Pilot Study: Establishing Glutamatergic Changes in Rapid Antidepressant Effects of Ketamine
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 857228
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Major Depressive Disorder (Experimental)
  Interventions: Drug: Ketamine only

INTERVENTIONS:
Drug: Ketamine only — The primary study intervention involves the administration of intravenous ketamine (0.5 mg/kg) over a 40-minute infusion. Ketamine, an NMDA receptor antagonist, has shown rapid antidepressant effects in individuals with treatment-resistant depression.

SUMMARY:
In the treatment of Major Depressive Disorder (MDD), ketamine can produce rapid but short-lasting improvements in mood. In order to develop a new generation of treatments with rapid and sustained efficacy, a better understanding of the mechanism of action is urgently needed. One candidate mechanism is the modulation of synaptic strength mediated by glutamatergic activity as ketamine has been suggested to increase synaptic strength. Although determining how ketamine impacts the glutamatergic system is essential to isolating its mechanism of action, the invasive nature of most assessment methods has limited our ability to do so in humans. The proposed research aims to determine if changes in glutamatergic activity, reflecting the modulation of synaptic strength, underlie the antidepressant effects of ketamine. In this project, the investigators will utilize a novel measure of glutamate imaging, GluCEST, to assess changes in glutamatergic activity to assess synaptic strength following ketamine administration. Ten individuals (aged 25-65) with a DSM-V diagnosis of MDD will undergo baseline GluCEST imaging prior to and following ketamine infusion. Both clinician-administered and subjective mood measures will be collected. It is predicted that ketamine will improve mood and increase glutamatergic activity and synaptic strength. Results from this project have the potential to identify the modifiable mechanisms by which rapid antidepressants work which could ultimately stimulate the development of novel interventions that work through the modulation of glutamatergic activity.

DETAILED DESCRIPTION:
Consent and Virtual Screening: Participants who meet initial inclusion criteria via phone screen will be invited to the complete a virtual visit that will include additional screening (e.g. Medical history), Structured Clinical Interview for DSMV (SCID) and clinician-administered measures of mood to determine final study eligibility. At the outset of this visit, all participants will receive verbal and written explanation of the general goals and risks of the study and will virtually sign an informed consent.

The results of the SCID will be used to characterize the study population and to determine whether they meet criteria for any diagnoses that would preclude participation (e.g. psychotic disorders). Their medical history will be reviewed by a study staff member to ensure that patients are diagnostically eligible.

At-home Sleep Recording: Following enrollment participants will complete a 7-day at-home sleep diary to assess sleep patterns prior to ketamine infusion. Sleep diaries will be completed either online via REDCap or with paper forms, based on participant preference and internet access.

In-laboratory Ketamine Infusion Protocol: On the study day, participants will arrive at the Hospital of the University of Pennsylvania at 9:00 AM. After initial orientation, they will undergo a baseline MRI scan between 9:00 AM and 11:00 AM. The MRI will utilize a 7T Siemens Terra system for high-resolution GluCEST imaging to capture glutamatergic activity. Following the scan, participants will complete baseline mood assessments, including the HAM-D, PANAS, VAS, and POMS scales. A light snack will be provided before the ketamine infusion begins between 12:00 PM and 1:00 PM. Participants will receive a 40-minute infusion of ketamine (0.5 mg/kg) under the supervision of a registered nurse and anesthesiologist. Continuous monitoring of vital signs (blood pressure, heart rate, oxygen levels) will be performed throughout the infusion. If adverse symptoms arise, the infusion may be paused or stopped at the discretion of the study physician. Following the infusion, participants will be observed for 1 hour to ensure stable vitals and recovery. Mood assessments will be repeated after the infusion to measure changes in emotional state. A second MRI scan will be conducted between 4:00 PM and 6:00 PM to assess changes in glutamatergic activity post-infusion. After completing the scan and final assessments, participants will be discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years;
2. Current depression as assessed on the SCID;
3. Treatment-resistant depression, as defined by failure of at least two previous antidepressant or mood stabilizing treatments within the current depressive episode. Failed antidepressant or mood stabilizing treatments can include pharmacotherapy for depression at an adequate dose for at least 8 weeks
4. Able to comprehend English, as all questionnaires are in this language
5. Ability to provide informed consent Ability to pass a comprehension assessment test related to effects of ketamine and trial objectives and criteria.

Exclusion Criteria:

1. A sleep disorder other than insomnia, as determined by history;
2. History of bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia and other psychotic disorders as assessed on the SCID;
3. Alcohol or drug abuse in the past year based upon the SCID or urine toxicology screen;
4. A current smoker;

4) Any significant medical or neurological illness that impacts brain function or impedes participation; 5) History of head trauma with significant loss of consciousness; 6) Metallic implants, pacemakers or tattoos, or other contraindications to MRI; Claustrophobic, or intolerant of the scanner environment; 7) For women, pregnancy will exclude participation. 8) Untreated hypertension

Based on ketamine's known difficulties with induction of perceptual/psychomimetic symptoms, exclusion criteria for this study are as follows:

1. Patients with a BMI over 40.
2. Ongoing prescription of 4 mg lorazepam equivalents (total) daily, or morning dosing of any benzodiazepine at the time of assessment;
3. Currently undergoing ECT, transcranial magnetic stimulation, vagal nerve stimulation, or deep brain stimulation as either an acute or maintenance treatment of depression;
4. Use of any MAOI is prohibited two weeks prior to administration of study drug; if patients are on an MAOI when enrolled, study drug will not be administered until two weeks off MAOI;
5. CYP3A4 inducers carbamazepine and modafinil are prohibited two weeks prior to administration of study drug and at least 24 hours after last dose of study drug.
6. Current use of Naltrexone;
7. Developmental delay, mental retardation, or intellectual disorder;
8. Clinical or self-reported diagnosis of delirium, encephalopathy, or related clinical diagnosis within the prior 12 months;
9. Prior participation in another study of ketamine for depression
10. Prior treatment and/or recreational use of ketamine

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
GluCEST imaging metrics | From pre to post-ketamine infusion (2 imaging sessions over a 9-hour span)
  relative change in glutamate concentration (% baseline)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | From pre to post-ketamine infusion (2 evaluations over a 9-hour span)
  Assessment of severity and change in depressive symptoms, from 0-52, with 52 indicating most severe

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Goldschmied, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No